CLINICAL TRIAL: NCT02087345
Title: Gastro-oesophageal Reflux in Oligosymptomatic Patients With Dental Erosion: a Longitudinal Study With pH-impedance Monitoring
Brief Title: Gastro-oesophageal Reflux in Oligosymptomatic Patients With Dental Erosion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brain-Gut Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: BGRG-2414b
Record Dates: First submitted 2014-03-10; First posted 2014-03-14 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Dental Erosion; Gastroesophageal Reflux
MeSH Terms: conditions — Tooth Erosion; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — gastric juice
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dental erosions

SUMMARY:
Dental erosions, the chemical dissolution of enamel without bacterial involvement, are considered to be an established complication of gastroesophageal reflux disease (GERD) by the Montreal global consensus statement. Given the high prevalence of dental erosions and the absence of any pH-impedance data or medical management guidelines for GERD-associated dental erosions, reflux characteristics will be characterized using questionnaires, endoscopy and esophageal pH-impedance testing, in successive patients dental erosions referred by dentists for evaluation of GERD. For assessment of the role of additional factors besides H+ activity in the refluxate, a sample of gastric juice will be aspirated during endoscopy and frozen for analysis of pepsin and other proteases. Prognostic factors for progression of dental erosions will be determined by repeating the evaluation after chronic dosing with esomeprazole 20mg twice-daily, which is prescribed to all patients.

ELIGIBILITY:
Inclusion criteria:

* Successive male and female patients
* Over 18 years of age presenting to the University of Bern Department of Dentistry and affiliated dentists
* Dental erosions

Exclusion criteria:

* Non-reflux causes of erosion
* Reduced salivary flow and buffering capacity
* History of bruxism, eating disorders, recurrent vomiting, severe obesity (BMI>35kg/m2) or past bariatric surgery
* Dietary or abrasive causes for dental erosion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Successive male and female patients with dental erosions
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-12-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The % of time with pH<4 and 5.5 during 24-hour pH-impedance | 1 year

SECONDARY OUTCOMES:
The number of acidic and weakly acidic reflux episodes during 24-hour pH-impedance | 1 year

OTHER OUTCOMES:
Association between dental erosion grades, gastric juice pepsin conc. and reflux episodes and % time with pH<4 and <5.5 during 24-hour pH-impedance | 1 year
  the % of reflux episodes reaching 15cm above the lower esophageal sphincter, concentration of pepsin and the tooth wear (BEWE) score: multivariate analysis with forward and backward elimination model to assess the best predicting variables.

CONTACTS AND LOCATIONS:
Overall Officials: Clive Wilder-Smith, MD, Principal Investigator — Brain-Gut Reserach Group
Locations (1):
- Gastroenterology Group Practice, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilder-Smith CH, Materna A, Martig L, Lussi A. Longitudinal study of gastroesophageal reflux and erosive tooth wear. BMC Gastroenterol. 2017 Oct 25;17(1):113. doi: 10.1186/s12876-017-0670-1. PMID 29070010